CLINICAL TRIAL: NCT02778711
Title: Anti-IL-17 a New Treatment for Contact Dermatititis
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tanja Todberg, MD (Other)
Responsible Party: Sponsor-Investigator, Tanja Todberg, MD, MD, University of Copenhagen
Organization: University of Copenhagen (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2015-004494-33
Record Dates: First submitted 2016-05-04; First posted 2016-05-20 (Estimated); Last update posted 2016-05-20 (Estimated); Status verified 2016-05

CONDITIONS: Allergic Contact Dermatitits
Keywords: anti-IL-17; secukinumab
MeSH Terms: interventions — secukinumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Cosentyx (Experimental): secukinumab (anti-IL-17)
  Interventions: Drug: secukinumab

INTERVENTIONS:
Drug: secukinumab — anti-IL-17
  Other Names: Cosentyx

SUMMARY:
The purpose of this study is to assess the efficacy of anti-IL 17 treatment (secukinumab) in patients with known severe allergic contact dermatitis (ACD).

DETAILED DESCRIPTION:
Purpose The purpose of this study is to assess the efficacy of anti-IL 17 treatment (secukinumab) in patients with known severe allergic contact dermatitis (ACD).

Background ACD is an immune mediated disease characterized by itching, erythema, vesicles, thickening and scaly skin, affecting a large part of the population in the world. A review study from 2007 by Thyssen et al that summarizes studies from North Europe and North America from 1966-2007 suggests that the prevalence to at least one allergen among these populations was 21.2 % (range 12.5-40.6%)(1). The incidence of ACD is not static and differs in countries(1), but in recent years there has been an increasing incidence of ACD caused by an increasing number of environmental detergents(2, 3). For patients with severe ACD the disease can be associated with difficulties performing daily activities, loss of sleep and reduced life quality (DLQI)(4).

ACD is treated with moisturizing creams, topical steroids and in severe cases systemic steroids, UVB, PUVA, azathioprin or alitretinoin. However, the drugs have severe side effects and some patients with ACD do not respond to the already existing treatments. New treatments are therefore highly needed. A group of these patients suffer from severe eczema often resulting in impared lifestyle and not seldom loss of work(4).

The pathogenesis in ACD is a T-cell mediated delayed type hypersensitivity reaction, consisting of a sensitization and an elicitation phase (5). In the sensitization phase an exogen allergen(hapten) is entering the epidermis through a defect skin barrier. The allergen is presented by the Langerhans cells to CD4+ and CD8+ T-cells in the lymphatic nodes, which activates and increases the numbers of T-cells. The elicitations phase begins when the patient once again is in contact with the allergen. The T-cells react with the allergen and this releases cytokines such as IFN-ɣ followed by skin lesions and inflammation. The IFN-ɣ is an important inflammatory cytokine, which is produced by CD4+ and CD8+ T-cells during ACD in humans and mice(6, 7). However, in the last decades studies have revealed that other inflammatory cytokines, such as IL-17 and IL-22 may be of importance in the immune response to contact allergens(8-11). IL-17 is produced by T-helper (TH)17 cells, innate cells as macrophages and dendrit cells and other cell types(12).

In mice both CD4+ and CD8+ T-cells producing IL-17 have been identified(13). A study by Nakae et al where IL-17 deficient mice were generated and exposed to dinitroflorobenzene and trinitrochlorobenzene, the mutants had a markedly reduced ear swelling compared to wild-type mice, this suggesting that IL-17 plays a role in contact allergy (14).

In nickel allergic humans, CD4+ and CD8+ T-cells have been shown to produce IL-17 and an increasing number of IL-17 producing cells have been found in tissue with eczematous reaction(8). Our group and others have found nickel-specific Th1 and Th17 cells in individuals with nickel allergy, but not in healthy controls(8, 9).

Our hypothesis is that since IL-17 appears to be involved in human ACD, anti-IL-17 treatment (secukinumab) might have a beneficial effect in patients with ACD.

This study will evaluate secukinumab treatment in patients with known allergic contact dermatitis. The study which is an interventional type will consist of two parts both performed at Department of Dermato-allergology, Herlev and Gentofte Hospital, University of Copenhagen, Hellerup, Denmark.

Study 1 Study 1 will include 10 patients with known allergy to nickel, but with no to low grade of eczema at inclusion.

Before enrollment patients will be screened for eligibility (blood samples (8-10 ml), Quantiferon TB Gold test, urine test for infection/pregnancy and chest x-ray to ensure that there is no evidence of infections and/or malignancy)(15).

The patients will then be tested with two standard patch tests with nickel and vehicle at the upper inner arm to confirm allergy. A photo and a biopsy (4 mm) from the patch test area will be taken, a clinical examination and a skinfold measure to evaluate the grade of dermatitis will be performed. The responses will be assessed clinically (at 48 h, 72 h and day 7) after application and graded as negative (-), doubtful (?+), 1+, 2+, 3+ or 4+ using a modified version of the International Contact Dermatitis Research (ICDRG) scoring system.

Patients will receive 300 mg secukinumab for s.c. injection (autoinjector) as a single dose, administered by a nurse at Department of Dermato-allergology, Gentofte Hospital. After one week the patients will be retested with nickel, photos and a biopsy from the patch test area will be taken, a clinical examination and a skinfold measure will be performed to evaluate the efficacy of secukinumab.

The study comprises 8 visits in total including screening

Study 2 Study 2 will include 10 patients with more than two known allergic contact allergies and clinically moderate to severe (PGA≥3) allergic contact dermatitis at inclusion. Patients will be treated open labeled for 8 weeks.

Before enrollment patients will be screened for eligibility (blood samples (20-25 ml), Quantiferon TB Gold test, urine test for infection/pregnancy and chest x-ray to ensure that there is no evidence of infections and/or malignancy)(15). Clinical degree of dermatitis will be evaluated by using Physician Global Assessment score (PGA) as an instrument for the severity of eczema with the following PGA levels: clear, almost clear, mild, moderate, severe. Dermatology Life Quality Index (DLQI, appendix 1) and Patient's Global Assessment score (PtGA, appendix 2) will be measured and photos of the eczema will be taken.

When test results from baseline clinical procedures are ready (7-14 days from screening visit) patients eligible for inclusion will have a biopsy taken (4 mm, at eczema), PGA, PtGA and DLQI will be performed and photos of eczema will be taken. This will be considered as baseline. Afterwards treatment with 300 mg secukinumab for s.c. injection (autoinjector) will initiate with the first dose administered by a nurse at Department of Dermato-allergology, Gentofte Hospital. During the first four weeks patients will be treated with secukinumab once a week. After this period secukinumab will be administered once a month with last dose given at week 8. All doses of secukinumab besides the first dose will be self-administered by the patients.

Two and four weeks from baseline another biopsy will be taken, PGA, PtGA and DLQI will be performed and photos of eczema will be taken to evaluate the efficacy of secukinumab. At week 4 another blood sample (12 ml) will be taken (cytokine level (IFN-ɣ and IL-17) will be evaluated) Eight and twelve weeks from baseline, PGA, PtGA and DLQI will be performed and photos will be taken to evaluate the efficacy of secukinumab. A follow up visit will be performed 16 weeks from baseline where relapse, PGA, PtGA, DLQI and safety during the treatment free weeks will be explored.

The study comprises 7 visits in total including screening

ELIGIBILITY:
Inclusion Criteria:

* Patients must be > 18
* Have a known nickel allergy with at least a +2 reaction when challenged with nickel
* Patients must have given their informed consent to the protocol and the clinical procedures
* Be able to speak and understand Danish.
* Patients must be > 18
* Have at least two known contact allergies
* Moderate to severe dermatitis at inclusion (PGA ≥ 3)
* Failure to local anti-inflammatory treatment and to at least one systemic anti-inflammatory treatment
* Patients must have given their informed consent to the protocol and the clinical procedures
* Be able to speak and understand Danish

Exclusion Criteria:

* Patients who have received any local anti-inflammatory treatment 2 weeks prior to day 0
* Patients who have received any systemic anti-inflammatory treatment 4 weeks prior to day 0
* Patients who have received any other study medication 4 weeks prior to day 0
* Dermatitis at the upper inner arm
* Patients with clinically significant disorders
* Patients with active TB/serious infections
* Pregnancy
* Nursing
* Women of child-bearing potential must use effective contraception which includes IUD, oral, injected or implanted hormonal device, hormone patch, vaginal hormonal ring, sterilization, occlusive cap or condom with spermicidal cream. Post-menopausal women (> 12 months of amenorrhea) are allowed not to use contraception.
* Patients who have received any weakened vaccines 6 weeks prior to day 0 or who are planning to receive a weakened vaccine during the study
* Latex allergy
* Patients who have received any local anti-inflammatory treatment 2 weeks prior to day 0
* Patients who have received any systemic anti-inflammatory treatment 4 weeks prior to day 0
* Patients who have received any other study medication 4 weeks prior to day 0
* Patients with clinically significant disorders
* Patients with active TB/serious infections
* Pregnancy
* Nursing
* Women of child-bearing potential must use effective contraception which includes IUD, oral, injected or implanted hormonal device, hormone patch, vaginal hormonal ring, sterilization, occlusive cap or condom with spermicidal cream. Post-menopausal women (> 12 months of amenorrhea) are allowed not to use contraception.
* Patients who have received any weakened vaccines 6 weeks prior to day 0 or who are planning to receive a weakened vaccine during the study
* Latex allergy

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2016-01; Primary Completion 2017-06 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
1. Reduction in clinical patch test score for dermatitis after secukinumab treatment compared to patch test score before treatment (study 1) | 18 months
Reduction in severity of eczema using the PGA score after treatment with secukinumab. | 18 months

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Dermato-Allergology, Hellerup, Denmark